CLINICAL TRIAL: NCT03797586
Title: Effect of Electroacupuncture on Opioid-induced Constipation in Patients With Cancer: Study Protocol for a Multicenter Randomized Controlled Trial
Brief Title: Effect of Electroacupuncture on Opioid-induced Constipation in Patients With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Liu Zhishun, Principal Investigator, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-164-KY-01
Record Dates: First submitted 2019-01-05; First posted 2019-01-09 (Actual); Results first posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Opioid-induced Constipation in Patients With Cancer
Keywords: electroacupuncture；opioid-induced constipation ,cancer

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electroacupuncture group (Experimental): Bilateral ST25,SP14, ST37 will be used in the EA group. For ST25 and SP14, 0.30×50mm or 0.30×75mm needles will be vertically inserted to the muscle layer of the abdominal , where patients will feel sharp pain and acupuncturists will feel resistance from the needle tip. For ST37, 0.30×40 mm needles will be vertically inserted approximately 15 mm deep, followed by three-time manipulation of even lifting and twisting method to elicit the sensation of deqi. Then paired alligator clips of the EA apparatus will be attached to the needle holders of the bilateral ST25, SP14, and ST37. EA stimulation will be retained for 30 minutes with a continuous wave of 10 Hz and current intensity of 0.5 to 4 mA.
  Interventions: Other: Electroacupuncture group
- Sham electroacupuncture group (Sham Comparator): Bilateral sham ST25, SP14, and ST37 will be used in the SA group. After sterilizing the skin, 0.30×40mm needles will be straightly inserted at the sham points about 2-3mm until they can be fixed on the skin when attached by the alligator clips. No manipulation will be used, and no deqi sensation are elicited for all sham points. The bilateral sham ST25, SP14, and ST37 points will be attached by the same EA apparatus with a continuous wave of 10 Hz and current intensity of 0.1 to 0.2 mA for 30 minutes with only the initial 30 seconds on.
  Interventions: Other: Sham electroacupuncture group

INTERVENTIONS:
Other: Electroacupuncture group — Bilateral Tianshu (ST25), Fujie (SP14), Shangjuxu (ST37) will be used in the EA group. With the local skin of the patients was routinely sterilized in a prone position in relaxation, acupuncturists will insert needles into the acupuncture points. For ST25 and SP14, 0.30×50mm or 0.30×75mm needles will be vertically inserted to the muscle layer of the abdominal wall, where participants will feel sharp pain and acupuncturists will feel resistance from the needle tip. For ST37, 0.30×40 mm needles will be vertically inserted approximately 15 mm deep, followed by three-time manipulation of even lifting and twisting method to elicit the sensation of deqi. Then paired alligator clips of the EA apparatus will be attached to the needle holders of the bilateral ST25, SP14, and ST37. EA stimulation will be retained for 30 minutes with a continuous wave of 10 Hz and current intensity of 0.5 to 4 mA.
  Arms: Electroacupuncture group
Other: Sham electroacupuncture group — Bilateral sham ST25, SP14, and ST37 will be used in the SA group. After sterilizing the skin, 0.30×40mm needles will be straightly inserted at the sham points about 2-3mm until they can be fixed on the skin when attached by the alligator clips. No manipulation will be used, and no deqi sensation are elicited for all sham points. The bilateral sham ST25, SP14, and ST37 points will be attached by the same EA apparatus with a continuous wave of 10 Hz and current intensity of 0.1 to 0.2 mA for 30 minutes with only the initial 30 seconds on.
  Arms: Sham electroacupuncture group

SUMMARY:
Approximately 70-80% of patients with advanced disease will be affected by moderate to severe pain. Opioid analgesics represented by morphine and oxycodone are the cornerstone of cancer-pain management, and recommended for use in the management of moderate to severe cancer pain according to WHO Cancer Pain Relief Guidelines. One view is that a trial of systemic opioid therapy should be administered to all cancer patients with pain of moderate or greater severity regardless of the pain mechanism. Although opioids analgesics do work well as relieving pain and improving quality of life via their action at opioid receptors in the central nervous system (CNS) and the peripheral nervous system, they also have powerful adverse effects. The overall occurrence of opioid-related adverse drug events has ranged from1.8% to 13.6%. Opioid-induced constipation (OIC), one of the most prevalent adverse events (AEs) in patients receiving opioid analgesics, defined as a change in baseline bowel habits or defecatory patterns following initiation, alteration, or increase in opioid therapy. The prevalence of OIC has been estimated to affect 41% of patients with chronic noncancer pain taking opioids and 94% of cancer patients taking opioids for pain. Unlike many other opioid-related AEs, OIC is persistent and rarely tolerated. OIC impacts pain control, patients' quality of life and may cause patients to reduce the dose or discontinue opioid use.

Acupuncture, a traditional Chinese medicine, has been used to treat gastrointestinal disease including constipation for thousands of years. Two systematic reviews concluded that acupuncture can improve spontaneous bowel movements for functional constipation, and our recent study indicated that electroacupuncture(EA) could increase complete spontaneous bowel movements and is safe for chronic severe functional constipation. Acupuncture could improve gastrointestinal function via facilitating gastrointestinal motility. Currently, there is little detailed information available regarding the acupuncture use for OIC. The objective of this study is to assess the efficacy and safety of EA for OIC in patients with cancer.

ELIGIBILITY:
Inclusion Criteria:

Cancer patients who conformed to all the following conditions will be further screened for eligibility:

1. Cancer patients must meet the Rome IV[1] diagnostic criteria for OIC: New or worsening symptoms of constipation following initiation, alteration, or increase in opioid treatment. For patients with a history of chronic functional constipation, he/she must have worsening symptoms of constipation when the opioid therapy is initiated, changed, or the dose is increased;
2. Patients recruited in this trial must have a history of OIC symptoms for at least 1 week;
3. Patients must be ≥18 years of age and ≤85 years of age;
4. Patient's cancer condition must be stable with a life expectancy that is more than six months;
5. Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-3;
6. Patients must have been receiving a relatively stable maintained opioid regimen, consisting of a total daily dose of 30 mg to 1000 mg oral morphine equivalents for at least 2 weeks prior to screening for cancer pain. Furthermore, it must be anticipated that the opioid will be maintained for at least 10 weeks;
7. The SBM frequency of the patients must be ≤ 2 times a week when laxatives are not being taken;
8. Patients must be capable of oral intake of drugs, food and beverages;
9. Provision of written informed consent before participation.

Exclusion Criteria:

Participants who fulfill any of the following criteria will be excluded:

1. Patients diagnosed with clinically significant abnormal defecation due to structural abnormalities of the gastrointestinal tract and other tissues related to gastrointestinal tract (not including OIC): inflammatory bowel disease, rectal prolapse, gastrointestinal obstruction, peritoneal metastasis, or peritoneal tumor at the time of enrollment;
2. Patients with a history of gastrointestinal tract operation, abdominal operation, or abdominal adhesion within one month prior to screening; history of intestinal obstruction within three months prior to screening;
3. Diagnosis of active diverticular disease; or severe hemorrhoid; or anal fissure; or artificial rectum or anus;
4. Patients with an intraperitoneal catheter or a feeding tube;
5. Diagnosis of pelvic disorder which are considered to have obvious effects on the intestinal transport of feces (such as uterine prolapse ≥degree 2, uterine fibroids [located in the posterior of the uterus with a diameter ≥ 5 cm] affecting bowel movement);
6. Patients that are being treated with a new cancer chemotherapy, which had never been administered in the past, within 14 days of the screening or are scheduled to receive such therapy during the study;
7. Patients that received radiotherapy within 28 days of the screening or are scheduled to receive such therapy during the study;
8. Patients that underwent a surgery or intervention that is considered to have an obvious effect on the gastrointestinal functions within 28 days of the screening or are scheduled to receive surgery or intervention which is considered to have obvious effects on the gastrointestinal functions during the study, or scheduled to receive surgery or intervention which will be anticipated to prevent the patients from completing the trial;
9. Patients with uncontrolled hyperthyroidism, severe hypertension, heart disease, systematic infection or blood coagulation disorders (hypercoagulation status or hemorrhagic tendency) at the time of study inclusion;
10. Patients that consumed >4 additional opioid doses per day, for breakthrough pain, for more than 3 days during the baseline period, or if their maintenance opioid dosing regimen was modified during this period;
11. Patients with severe cancerous pain (e.g., typical average daily pain intensity rating of 7 to 10 on a numerical rating scales (NRS; 0 [no pain] to 10 [the worst pain possible]) after the use of routine dose and frequency of opioids) refractory to opioid therapy;
12. Patients with a history of opioid discontinuation due to severe adverse events or patients that are expected to discontinue opioid use due to the potential risk of adverse events;
13. Patients that received an opioid receptor antagonist within one month of the screening, or those who are scheduled to receive such therapy during the study;
14. Patients with a history of nerve neurolysis;
15. Patients with severe cognitive impairment, aphasia, or psychiatric disorders; abdominal aortic aneurysm; hepatomegaly(liver span > 14cm at the mid-clavicular line by ultrasound examination); or splenomegaly (spleen length [cranial to caudal] > 13cm by ultrasound examination);
16. Patients that have received acupuncture within three months of the screening;
17. Other patients who are considered ineligible for the study by the investigator on the basis of concomitant therapy and medical findings.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-10-16 (Actual); Study Completion 2021-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhishun Liu, Study Chair — China Academy of Chinese Medicine Sciences
Locations (1):
- Guang An Men Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang W, Liu Y, Yang X, Sun J, Yue Z, Lu D, Zhou K, Sun Y, Hou A, Zang Z, Jin X, Liu C, Wang Y, Yu J, Zhu L, Liu Z. Effects of Electroacupuncture for Opioid-Induced Constipation in Patients With Cancer in China: A Randomized Clinical Trial. JAMA Netw Open. 2023 Feb 1;6(2):e230310. doi: 10.1001/jamanetworkopen.2023.0310. PMID 36811861
- [Derived] Wang W, Wang X, Liu Y, Sun Y, Liu X, Yan Y, Liu Z. Effects of Electroacupuncture on Opioid-Induced Constipation in Patients With Cancer: Study Protocol for a Multicenter Randomized Controlled Trial. Front Med (Lausanne). 2022 Apr 13;9:818258. doi: 10.3389/fmed.2022.818258. eCollection 2022. PMID 35492306

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Electroacupuncture Group | Sham Electroacupuncture Group
Started | 50 | 50
Completed | 46 | 41
Not Completed | 4 | 9
Not completed — Lost to Follow-up | 3 | 6
Not completed — Death | 1 | 1
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Electroacupuncture Group: Bilateral Tianshu (ST25), Fujie (SP14), Shangjuxu (ST37) will be used in the EA group. The location of the acupoints will be based on Nomenclature and location of acupuncture points34 drafted in 2006 by the National Standard of the People's Republic of China (GB/T 12346-2006). The local skin will be routinely sterilized while the patient is in a supine position. For ST25 and SP14, 0.30×50 mm or 0.30×75 mm needles will be gently vertically inserted to the muscle layer of the abdominal wall, where patients will feel sharp pain and acupuncturists will feel resistance from the needle tip. For ST37, 0.30×40 mm needles will be vertically inserted approximately 15 mm deep, followed by three-time manipulation of even lifting and twisting method to elicit the sensation of deqi. Paired alligator clips of the EA apparatus will then be attached to the needle holders of the bilateral ST25, SP14, and ST37. The stimulation will be retained for 30 minutes, with a continuous wave of 10 Hz and current intensity of 0.5 to 4 mA. All needles will be removed after 30 minutes and pressure will be applied using a dry sterilized cotton ball to avoid bleeding. Patients will receive 24 treatment sessions over an 8-week period (3 sessions each week, ideally every other day). Patients will be followed up for another 8 weeks after the treatment stopped.
- Sham Electroacupuncture Group: The patients in the sham electroacupuncture group will receive minimal needling at non-acupoints as bilateral sham ST25, SP14, and ST37. The sham ST25 and SP14 are located 2 cm horizontally outward of the points stimulaed in the EA group. The sham ST37 point is located outward of ST37 in the middle of the stomach and gallbladder channel. After sterilization of the skin, 0.30×40 mm needles will be directly inserted about 2-3 mm until they can stand up when attached by the alligator clips. No manipulation will be used and no deqi sensation will be elicited at any of the sham points. The bilateral sham ST25, SP14, and ST37 points will be attached by the same EA apparatus with a continuous wave of 10 Hz and current intensity of 0.1 to 0.2 mA for 30 minutes with only the initial 30 seconds on. Patients will receive 24 treatment sessions over an 8-week period (3 sessions each week, ideally every other day). Patients will be followed up for another 8 weeks after the treatment stopped.
- Total: Total of all reporting groups
Arm/Group | Electroacupuncture Group | Sham Electroacupuncture Group | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.60 (10.40) | 65.12 (10.64) | 64.36 (10.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 23 | 44
  Male | 29 | 27 | 56
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Han | 48 | 49 | 97
  Others | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  China | 50 | 50 | 100
ECOG performance status [Count of Participants; unit: Participants] — Values for ECOG performance status range from 0 to 5; higher scores indicate greater disability.
  Participants
    0 | 0 | 1 | 1
    1 | 3 | 7 | 10
    2 | 36 | 22 | 58
    3 | 11 | 20 | 31
Type of primary cancer [Count of Participants; unit: Participants]
  Lung | 17 | 21 | 38
  Breast | 5 | 3 | 8
  Colorectal | 2 | 1 | 3
  Stomach | 2 | 1 | 3
  Others | 24 | 24 | 48
Patients with cancer metastasis upon enrollment [Count of Participants; unit: Participants] | 21 | 27 | 48
Type of treatment received at baseline [Count of Participants; unit: Participants]
  Radiotherapy | 3 | 8 | 11
  Chemotherapy | 33 | 19 | 52
  Chemotherapy + radiotherapy | 5 | 8 | 13
  Targeted therapy | 7 | 11 | 18
  Other | 2 | 4 | 6
Type of opioid administered [Count of Participants; unit: Participants]
  Oxycodone | 25 | 39 | 64
  Morphine | 10 | 6 | 16
  Others | 15 | 5 | 20
No. of patients stratified by opioid dose [Count of Participants; unit: Participants]
  30-100 mg | 37 | 38 | 75
  >100 mg | 13 | 12 | 25
History of chronic functional constipation [Count of Participants; unit: Participants] | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Response
Description: A responder（Participant With Response） is defined as a patient that has at least three spontaneous bowel movements (SBMs) per week and an increase of at least one SBM a week from the baseline for at least 6 of the 8 weeks of the treatment period.
Time Frame: weeks 1-8
Population: Three participants in the electroacupuncture group and 5 participants in the sham electroacupuncture group did not complete 8-week treatment over weeks 1-8.
Measure: Number; unit: participants
Arm/Group | Electroacupuncture Group | Sham Electroacupuncture Group
Number analyzed (Participants) | 47 | 45
participants | 19 | 4

2. Secondary Outcome: A Change in the Mean Weekly Spontaneous Bowel Movements (SBMs) From the Baseline During Weeks 1-8 and Weeks 13-16.
Description: An SBM was defined as a bowel movement that occurred without any medication or intervention to assist defection within the previous 24 hours. A bowel movement occurring within 24 hours of an optional assisted method for defecation was not considered to be an SBM. The mean weekly spontaneous bowel movements (SBMs) during weeks 1-8 and weeks 13-16 is calculated by dividing the total frequency of SBMs by the number of weeks recorded.
Time Frame: weeks 1-8, and weeks 13-16
Population: Three participants in the electroacupuncture group and 5 participants in the sham electroacupuncture group did not complete 8-week treatment over weeks 1-8. One participant in the electroacupuncture group and 4 participants in sham electroacupuncture group dropped out over weeks 9-16.
Measure: Mean (95% Confidence Interval); unit: spontaneous bowel movements/week
Arm/Group | Electroacupuncture Group | Sham Electroacupuncture Group
Number analyzed (Participants) | 47 | 45
spontaneous bowel movements/week
  weeks 1-8 | 1.17 [1 to 1.34] | 0.61 [0.43 to 0.78]
  weeks 13-16: number analyzed (Participants) | 46 | 41
  weeks 13-16 | 0.59 [0.42 to 0.78] | 0.23 [0.04 to 0.43]

3. Secondary Outcome: Number of Participants With ≥3 Mean Weekly Spontaneous Bowel Movements (SBMs) During Weeks 1-8
Description: An SBM was defined as a bowel movement that occurred without any medication or intervention to assist defection within the previous 24 hours. A bowel movement occurring within 24 hours of an optional assisted method for defecation was not considered to be an SBM. The mean weekly spontaneous bowel movements (SBMs) during weeks 1-8 is calculated by dividing the total frequency of SBMs by the number of weeks recorded.
Time Frame: weeks 1-8
Measure: Count of Participants; unit: Participants
Arm/Group | Electroacupuncture Group | Sham Electroacupuncture Group
Number analyzed (Participants) | 47 | 45
Participants | 19 | 6

4. Secondary Outcome: Number of Participants With ≥3 Mean Weekly Spontaneous Bowel Movements (SBMs) During Weeks 13-16
Description: An SBM was defined as a bowel movement that occurred without any medication or intervention to assist defection within the previous 24 hours. A bowel movement occurring within 24 hours of an optional assisted method for defecation was not considered to be an SBM.The mean weekly spontaneous bowel movements (SBMs) during weeks 13-16 is calculated by dividing the total frequency of SBMs by the number of weeks recorded.
Time Frame: weeks 13-16
Measure: Count of Participants; unit: Participants
Arm/Group | Electroacupuncture Group | Sham Electroacupuncture Group
Number analyzed (Participants) | 46 | 41
Participants | 4 | 1

5. Secondary Outcome: Number of Participants With an Increase of ≥1 Mean Weekly Spontaneous Bowel Movements (SBMs) From the Baseline During Weeks 1-8
Description: as for outcome 3
Time Frame: weeks 1-8
Measure: Count of Participants; unit: Participants
Arm/Group | Electroacupuncture Group | Sham Electroacupuncture Group
Number analyzed (Participants) | 47 | 45
Participants | 30 | 14

6. Secondary Outcome: Number of Participants With an Increase of ≥1 Mean Weekly Spontaneous Bowel Movements (SBMs) From the Baseline During Weeks 13-16
Description: An SBM was defined as a bowel movement that occurred without any medication or intervention to assist defection within the previous 24 hours. A bowel movement occurring within 24 hours of an optional assisted method for defecation was not considered to be an SBM. The mean weekly spontaneous bowel movements (SBMs) during weeks 13-16 is calculated by dividing the total frequency of SBMs by the number of weeks recorded.
Time Frame: weeks 13-16
Measure: Count of Participants; unit: Participants
Arm/Group | Electroacupuncture Group | Sham Electroacupuncture Group
Number analyzed (Participants) | 46 | 41
Participants | 12 | 4

7. Secondary Outcome: A Change in the Mean Weekly Complete Spontaneous Bowel Movements (CSBMs) From the Baseline During Weeks 1-8 and Weeks 13-16.
Description: An SBM was defined as a bowel movement that occurred without any medication or intervention to assist defection within the previous 24 hours. A bowel movement occurring within 24 hours of an optional assisted method for defecation was not considered to be an SBM. A CSBM was defined as an SBM with the feeling of complete evacuation. The mean weekly complete spontaneous bowel movements (CSBMs) during weeks 1-8 and weeks 13-16 is calculated by dividing the total frequency of CSBMs by the number of weeks recorded.
Time Frame: weeks 1-8, and weeks 13-16
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: CSBMs/week
Arm/Group | Electroacupuncture Group | Sham Electroacupuncture Group
Number analyzed (Participants) | 47 | 45
CSBMs/week
  Week 1-8 | 0.84 [0.65 to 1.02] | 0.35 [0.16 to 0.54]
  Week 13-16: number analyzed (Participants) | 46 | 41
  Week 13-16 | 0.32 [0.14 to 0.51] | 0.14 [-0.06 to 0.33]

8. Secondary Outcome: Number of Participants With ≥3 Mean Weekly Spontaneous Bowel Movements (CSBMs) During Weeks 1-8
Description: An SBM was defined as a bowel movement that occurred without any medication or intervention to assist defection within the previous 24 hours. A bowel movement occurring within 24 hours of an optional assisted method for defecation was not considered to be an SBM. A CSBM was defined as an SBM with the feeling of complete evacuation.
Time Frame: weeks 1-8
Measure: Count of Participants; unit: Participants
Arm/Group | Electroacupuncture Group | Sham Electroacupuncture Group
Number analyzed (Participants) | 47 | 45
Participants | 0 | 0

9. Secondary Outcome: Number of Participants With ≥3 Mean Weekly Spontaneous Bowel Movements (CSBMs) During Weeks 13-16
Description: as for outcome 8
Time Frame: weeks 13-16
Measure: Count of Participants; unit: Participants
Arm/Group | Electroacupuncture Group | Sham Electroacupuncture Group
Number analyzed (Participants) | 46 | 41
Participants | 1 | 0

10. Secondary Outcome: Number of Participants With an Increase of ≥1 Mean Weekly Spontaneous Bowel Movements (CSBMs) From the Baseline During Weeks 1-8
Description: as for outcome 8
Time Frame: weeks 1-8
Measure: Count of Participants; unit: Participants
Arm/Group | Electroacupuncture Group | Sham Electroacupuncture Group
Number analyzed (Participants) | 47 | 45
Participants | 21 | 9

11. Secondary Outcome: Number of Participants With an Increase of ≥1 Mean Weekly Spontaneous Bowel Movements (CSBMs) From the Baseline During Weeks 13-16
Description: as for outcome 8
Time Frame: weeks 13-16
Measure: Count of Participants; unit: Participants
Arm/Group | Electroacupuncture Group | Sham Electroacupuncture Group
Number analyzed (Participants) | 46 | 41
Participants | 10 | 4

12. Secondary Outcome: A Change in the Mean Bristol Stool Form Scale Score for Stool Consistency of Spontaneous Bowel Movements (SBMs) From the Baseline During Weeks 1-8 and Weeks 13-16
Description: For stool consistency, each patient was asked to record their stool consistency according to the Bristol Stool Form Scale, on the following seven points scale (scored from 1 to 7 for stool types 1 to 7, respectively) .Higher scores indicate indicating a softer stool.The mean Bristol Stool Form Scale score for stool consistency of spontaneous bowel movements (SBMs) during weeks 1-8 and weeks 13-16 is calculated by dividing the total Bristol Stool Form Scale score of SBMs by the total number of SBMs recorded.
Time Frame: weeks 1-8, and weeks 13-16
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Electroacupuncture Group | Sham Electroacupuncture Group
Number analyzed (Participants) | 47 | 45
score on a scale
  Week 1-8 | 0.51 [0.29 to 0.73] | 0.28 [0.05 to 0.50]
  Week 13-16: number analyzed (Participants) | 46 | 41
  Week 13-16 | 0.25 [0.01 to 0.49] | -0.07 [-0.32 to 0.18]

13. Secondary Outcome: A Change in the Mean Score for the Straining of Spontaneous Bowel Movements (SBMs) From the Baseline During Weeks 1-8 and Weeks 13-16
Description: For assessment of straining of spontaneous bowel movement (SBM), each patient was asked to rate his/her score for straining using the following five-point scale: not at all difficulty (0), a little bit difficulty (1), moderately difficulty (2), quite a bit difficulty (3), extremely difficulty (4). Higher scores indicate a worse outcome.The mean score for the straining of SBMs during weeks 1-8 and weeks 13-16 is calculated by dividing the total score for the straining of SBMs by the total number of SBMs recorded.
Time Frame: weeks 1-8, and weeks 13-16
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Electroacupuncture Group | Sham Electroacupuncture Group
Number analyzed (Participants) | 47 | 45
score on a scale
  Weeks 1-8 | -0.58 [-0.78 to -0.39] | -0.12 [-0.32 to 0.08]
  Weeks 13-16: number analyzed (Participants) | 46 | 41
  Weeks 13-16 | -0.30 [-0.52 to -0.08] | 0.04 [-0.19 to 0.27]

14. Secondary Outcome: A Change in the Total Score of the Patient Assessment of Constipation-Symptom (PAC-SYM) Questionnaire From Baseline at Weeks 8 and 16
Description: The Patient Assessment of Constipation-Symptom (PAC-SYM) is a 12-item evaluative questionnaire for the chronic constipation, which consists of 4-item abdominal, 3-item rectal, and 5-item stool subscales. Each item score ranges from 0 to 4 in the 2 weeks (14 days) prior to assessment，where 0 = symptom absent, 1 = mild,2 = moderate,3 = severe and 4 = very severe. Each subscale score will be calculated as the mean of the completed items for that subscale，which will range from 0 to 4. The total score will be calculated as the mean of all subscales. The total score of PAC-SYM range from 0 to 4.Lower scores indicate a better outcome. The specific evaluation of total scores of the PAC-SYM occurs at both week 8 and week 16.
Time Frame: week 8 and week 16
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Electroacupuncture Group | Sham Electroacupuncture Group
Number analyzed (Participants) | 47 | 45
score on a scale
  Week 8 | -0.87 [-1.01 to -0.73] | -0.51 [-0.65 to -0.37]
  Week 16: number analyzed (Participants) | 46 | 41
  Week 16 | -0.47 [-0.61 to -0.33] | -0.11 [-0.27 to 0.04]

15. Secondary Outcome: A Change in the Total Scores of the Patient Assessment of Constipation-Quality of Life (PAC-QOL) Questionnaires From the Baseline at Weeks 8 and 16
Description: The Patient Assessment of Constipation-Quality of Life (PAC-QOL) is a 28-item self-reported instrument for assessing the burden of constipation on patients' everyday functioning and well-being in the 2 weeks (14 days) prior to assessment. It is divided into four subscales: physical discomfort (items 1-4), psychosocial discomfort (items 5-12), worries/concerns (items 13-23), and satisfaction (items 24 to 28). Each of the item scores ranges from 0 (not at all) to 4 (extremely). Each of the item scores ranges from 0 (not at all) to 4 (extremely), with lower scores indicating a better quality of life. The each subscale score ranges from 0 to 4. The total score will be calculated as the mean of all subscales, ranging from 0 to 4. Lower scores indicate a better outcome. The specific evaluation of the PAC-QOL questionnaires' total scores occurs at both week 8 and week 16.
Time Frame: week 8 and week 16
Population: as for outcome 2
Measure: Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | Electroacupuncture Group | Sham Electroacupuncture Group
Number analyzed (Participants) | 47 | 45
units on a scale
  Week 8 | -0.62 [-0.76 to -0.48] | -0.36 [-0.51 to -0.22]
  Week 16: number analyzed (Participants) | 46 | 41
  Week 16 | -0.36 [-0.53 to -0.20] | -0.11 [-0.27 to 0.06]

16. Secondary Outcome: Patients'Global Assessment of Treatment Efficacy
Description: Each patient was asked to rate his/her efficacy of treatment using the following 7-point self-reporting scale: markedly worse (1), moderately worse (2),slightly worse (3), no change (4), slightly improved (5), moderately improved (6), markedly improved (7). Higher scores mean a better outcome.
Time Frame: week 8 and week 16
Population: Three participants in the electroacupuncture group and 5 participants in the sham electroacupuncture group in week 8. Four participants in the electroacupuncture group and 9 participants in the sham electroacupuncture group in week 16.
Measure: Count of Participants; unit: Participants
Arm/Group | Electroacupuncture Group | Sham Electroacupuncture Group
Number analyzed (Participants) | 47 | 45
Participants
  Week 8: Markedly improved | 13 | 3
  Week 8: Moderately improved | 21 | 4
  Week 8: Slightly improved | 10 | 30
  Week 8: No change | 2 | 8
  Week 8: Slightly worse | 0 | 0
  Week 8: Moderately worse | 1 | 0
  Week 8: Markedly worse | 0 | 0
  Week 16: number analyzed (Participants) | 46 | 41
  Week 16: Markedly improved | 8 | 0
  Week 16: Moderately improved | 6 | 1
  Week 16: Slightly improved | 13 | 10
  Week 16: No change | 3 | 19
  Week 16: Slightly worse | 6 | 1
  Week 16: Moderately worse | 6 | 5
  Week 16: Markedly worse | 4 | 5

17. Secondary Outcome: Number of Participants Using Rescue Medicine During Weeks 1-8 and Weeks 9-16
Description: The percentage of patients using rescue medicine will be compared between groups during weeks 1-8, and weeks 9-16. The mean frequency of using rescue medicine per week during weeks 1-8 equals the total of rescue medicine consumption divided by 8. The mean frequency of using rescue medicine per week during weeks 9-16 equals the total of rescue medicine consumption divided by 8.
Time Frame: weeks 1-8, and weeks 9-16
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Electroacupuncture Group | Sham Electroacupuncture Group
Number analyzed (Participants) | 47 | 45
participants
  Weeks 1-8 : Rescue medicine | 24 | 30
  Weeks 1-8 : Others | 5 | 4
  Weeks 9-16 : Rescue medicine: number analyzed (Participants) | 46 | 41
  Weeks 9-16 : Rescue medicine | 28 | 29
  Weeks 9-16 : Others: number analyzed (Participants) | 46 | 41
  Weeks 9-16 : Others | 5 | 2

18. Secondary Outcome: The Mean Frequency of Rescue Medicine Use Per Week During Weeks 1-8 and Weeks 9-16
Description: The mean frequency of using rescue medicine per week during weeks 1-8 equals the total of rescue medicine consumption divided by 8. The mean frequency of using rescue medicine per week during weeks 9-16 equals the total of rescue medicine consumption divided by 8.
Time Frame: weeks 1-8, and weeks 9-16
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: number of rescue medicine use per week
Arm/Group | Electroacupuncture Group | Sham Electroacupuncture Group
Number analyzed (Participants) | 47 | 45
number of rescue medicine use per week
  Weeks 1-8 : Rescue medicine | 0.39 [0.2 to 0.59] | 0.65 [0.48 to 0.82]
  Weeks 1-8 : Others | 0.70 [0.15 to 1.25] | 0.94 [0.34 to 1.54]
  Weeks 9-16 : Rescue medicine: number analyzed (Participants) | 46 | 41
  Weeks 9-16 : Rescue medicine | 0.62 [0.42 to 0.82] | 0.85 [0.66 to 1.05]
  Weeks 9-16 : Others: number analyzed (Participants) | 46 | 41
  Weeks 9-16 : Others | 0.46 [-0.05 to 0.97] | 0.47 [-0.38 to 1.31]

19. Other Pre Specified Outcome: Patients'Expectation of the Acupuncture Efficacy
Description: Participants will be asked to answer the following questions before the intervention: "Do you think acupuncture will be effective in treating the disease in general?" "Do you think acupuncture will be effective in improving the OIC?" and "which acupuncture modalities do you prefer, EA or SA?" For each question, patients will choose one of the following answers: "unclear/whatever", "EA", or "SA"
Time Frame: at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Electroacupuncture Group | Sham Electroacupuncture Group
Number analyzed (Participants) | 50 | 50
Participants
  Do you think acupuncture will be effective in treating diseases in general?: Yes | 38 | 35
  Do you think acupuncture will be effective in treating diseases in general?: No | 0 | 0
  Do you think acupuncture will be effective in treating diseases in general?: Unclear | 12 | 15
  Do you think acupuncture will be effective for opioid-induced constipation?: Yes | 31 | 29
  Do you think acupuncture will be effective for opioid-induced constipation?: No | 0 | 0
  Do you think acupuncture will be effective for opioid-induced constipation?: Unclear | 19 | 21

20. Other Pre Specified Outcome: The Patient Blinding Assessment
Description: Before treatment, we told participants that they had a 50% chance of receiving conventional electroacupuncture with a deeper insertion or minimal electroacupuncture with a superficial penetration. Conventional electroacupuncture and minimal electroacupuncture have probable similar efficacy. Both treatmentsused a relatively small electric intensity, and they may or may not feel the stimulation during treatment because of the relatively weak electrical stimulation and the tolerance of the human body. To assess the success of blinding, within 5 minutes after any treatment session at week 8, participants were asked to guess whether they had received conventional electroacupuncture in the previous weeks (yes or no)
Time Frame: at week 8
Population: Answers from 3 participant in the electroacupuncture group and 5 participants in the sham electroacupuncture group were not recorded due to staff negligence.
Measure: Count of Participants; unit: Participants
Arm/Group | Electroacupuncture Group | Sham Electroacupuncture Group
Number analyzed (Participants) | 47 | 45
Participants
  Guess Conventional electroacupuncture | 46 | 22
  Guess Minimal electroacupuncture | 1 | 23

21. Other Pre Specified Outcome: Change in Numeric Rating Scales Score for Mean Cancer Pain Intensity Within the Preceding Week From Baseline
Description: The mean cancerous pain intensity and worst cancerous pain intensity during the preceding week will be evaluated by 11 grades (from "0=no pain" to "10=worst pain (the strongest pain ever experienced)" at baseline, as well as weeks 2, 4, 6, 8 and 16. Higher scores mean a worse outcome. The values at weeks 2, 4, 6, and 8 are summed and divided by 4. Value at week 16 is a single value.
Time Frame: at baseline, at weeks 8 and 16.
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Electroacupuncture Group | Sham Electroacupuncture Group
Number analyzed (Participants) | 47 | 45
score on a scale
  Week 8 | -0.17 [-0.36 to 0.01] | -0.003 [-0.19 to 0.19]
  Week 16: number analyzed (Participants) | 46 | 41
  Week 16 | -0.09 [-0.37 to 0.20] | 0.14 [-0.15 to 0.44]

22. Other Pre Specified Outcome: Change in Numeric Rating Scales Score for Worst Cancer Pain Intensity Within the Preceding Week From Baseline
Description: The mean cancerous pain intensity and worst cancerous pain intensity during the preceding week will be evaluated by 11 grades (from "0=no pain" to "10=worst pain (the strongest pain ever experienced)" at baseline, as well as weeks 2, 4, 6, 8 and 16. Higher scores mean a worse outcome.The values at weeks 2, 4, 6, and 8 are summed and divided by 4. Value at week 16 is a single value.
Time Frame: at baseline, at weeks 8 and 16.
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Electroacupuncture Group | Sham Electroacupuncture Group
Number analyzed (Participants) | 47 | 45
score on a scale
  Week 8 | -0.19 [-0.44 to 0.05] | -0.07 [-0.32 to 0.18]
  Week 16: number analyzed (Participants) | 46 | 41
  Week 16 | 0.03 [-0.35 to 0.42] | 0.23 [-0.17 to 0.63]

23. Other Pre Specified Outcome: Number of Participants With Change From Baseline in the Dose of Opioid Consumption From Baseline During Weeks 1-8
Description: The percentage of patients discontinuing the opioid, and those with increase/decrease from baseline of ≥30% opioid usage per week was compared between groups during weeks 1-8
Time Frame: at week 8
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Electroacupuncture Group | Sham Electroacupuncture Group
Number analyzed (Participants) | 47 | 45
participants
  Remained unchanged | 40 | 34
  Participants with the opioid consumption increase ≥30% | 6 | 7
  Participants with the opioid consumption increase <30% | 1 | 4
  Participants with the opioid consumption decrease ≥30% | 0 | 0
  Participants with the opioid consumption decrease <30% | 0 | 0

24. Other Pre Specified Outcome: Number of Participants With Change From Baseline in the Dose of Opioid Consumption From Baseline During Weeks 9-16
Description: The percentage of patients discontinuing the opioid, and those with increase/decrease from baseline of ≥30% opioid usage per week was compared between groups during weeks 9-16
Time Frame: at week 16
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Electroacupuncture Group | Sham Electroacupuncture Group
Number analyzed (Participants) | 46 | 41
participants
  Remained unchanged | 33 | 29
  Participants with the opioid consumption increase ≥30% | 10 | 9
  Participants with the opioid consumption increase <30% | 3 | 3
  Participants with the opioid consumption decrease ≥30% | 0 | 0
  Participants with the opioid consumption decrease <30% | 0 | 0

25. Post Hoc Outcome: Number of Participants With Sustained SBM(Spontaneous Bowel Movements) Response
Description: Responders are defined as those having at least three SBMs per week and an increase from baseline of at least one SBM per week for at least 6 weeks out of the 8-week treatment period. The percentage of sustained SBM(spontaneous bowel movements) responders is defined as patients who fulfilled these criteria for at least 3 of the last 4 weeks'treatment.
Time Frame: over weeks 1-8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Electroacupuncture Group | Sham Electroacupuncture Group
Number analyzed (Participants) | 47 | 45
Participants | 19 | 4

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) will be recorded throughout the whole trial(17 weeks) in Adverse Event Form (AEF) by patients themselves and outcome assessors.
Arm/Group | Electroacupuncture Group | Sham Electroacupuncture Group
All-Cause Mortality (participants affected / at risk) | 1/50 | 1/50
Serious Adverse Events (participants affected / at risk) | 1/50 | 3/50
Other Adverse Events (participants affected / at risk) | 3/50 | 5/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Electroacupuncture Group (N=50) | Sham Electroacupuncture Group (N=50)
Death (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Death was due to lung cancer. It was considered not related to acupuncture treatment by the investigator.
Death (Immune system disorders) | 0 (0) | 1 (1) — Death was due to malignant lymphoma. It was considered not related to acupuncture treatment by the investigator.
Cancer progression (Immune system disorders) | 0 (0) | 1 (1) — Cancer progression was due to the preexisting condition. It was considered not related to acupuncture treatment by the investigator.
Cancer progression (Reproductive system and breast disorders) | 0 (0) | 1 (1) — Cancer progression was due to the preexisting condition. It was considered not related to acupuncture treatment by the investigator.
OTHER ADVERSE EVENTS (reported when occurring in more than 0.02% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Electroacupuncture Group (N=50) | Sham Electroacupuncture Group (N=50)
Local hematoma (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
Inconsequential bleeding (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2019-11-29): https://cdn.clinicaltrials.gov/large-docs/86/NCT03797586/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2021-12-10): https://cdn.clinicaltrials.gov/large-docs/86/NCT03797586/SAP_001.pdf